CLINICAL TRIAL: NCT01158729
Title: Antithrombin III Supplementation Prior to Cardiopulmonary Bypass for Neonates
Brief Title: Antithrombin III Supplementation for Cardiopulmonary Bypass in Neonates
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Grant funding expired, poor patient enrollment
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's National Research Institute (Other); rEVO Biologics (Industry)
Responsible Party: Principal Investigator, Robert Niebler, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ped-ATIII CPB 001
Record Dates: First submitted 2010-06-17; First posted 2010-07-08 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Postoperative Hemorrhage
Keywords: Antithrombin III; Postoperative Hemorrhage; Cardiopulmonary Bypass; Pediatrics; Blood Transfusion
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Antithrombins; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATIII experimental group (Experimental): 30 neonates (4-30 days of age) undergoing surgery requiring cardiopulmonary bypass will receive Antithrombin (Recombinant) prior to initiation of bypass
  Interventions: Drug: Antithrombin (Recombinant)
- Placebo Controls (Placebo Comparator): 30 neonates (4-30 days of age) undergoing surgery requiring cardiopulmonary bypass will receive placebo prior to initiation of bypass
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Antithrombin (Recombinant) — Single dose of antithrombin (recombinant) to be given prior to initiation of cardiopulmonary bypass. Intravenous dose determined by following formula: ATIII dose given to patient = [(1.0 Units/mL - patient's measured ATIII concentration in Units/mL) X weight (kg) X 80 mL/kg] X (1 mL/175 Units)
  Other Names: ATryn; Recombinant antithrombin
  Arms: ATIII experimental group
Other: Placebo — Single dose of placebo (0.9% NaCl) to be given prior to initiation of cardiopulmonary bypass. Intravenous dose determined by following formula: Placebo dose given to patient = [(1.0 Units/mL - patient's measured ATIII concentration in Units/mL) X weight (kg) X 80 mL/kg] X (1 mL/175 Units)
  Other Names: 0.9% NaCl; Normal Saline
  Arms: Placebo Controls

SUMMARY:
A prospective, randomized, placebo-controlled, double-blinded pilot study is planned. Neonates undergoing surgeries requiring cardiopulmonary bypass will receive antithrombin III (ATIII) supplementation or placebo in addition to standard anticoagulation with heparin as currently practiced at Children's Hospital of Wisconsin. We plan to enroll the first 60 sequential patients meeting criteria who consent to inclusion. The primary outcomes will be rates of adverse events to monitor safety. Secondary outcomes include volume of postoperative blood loss and packed red blood cell transfusion during the first 24 postoperative hours, and ATIII levels during and after bypass to determine pharmacokinetics.

DETAILED DESCRIPTION:
Hypothesis:

ATIII supplementation prior to initiation of cardiopulmonary bypass (CPB) to neonates will be safe and result in less postoperative bleeding and transfusion of packed red blood cells (pRBC) as compared to placebo controls.

Specific Aims:

1. To determine the safety and feasibility of ATIII supplementation prior to initiation of CPB in neonates.
2. To determine the pharmacokinetics of ATIII supplementation prior to initiation of CPB in neonates
3. To compare the postoperative blood loss and pRBC transfusion requirements in an experimental group of neonates undergoing surgery requiring CPB who receive ATIII prior to initiation of CPB to that of a placebo control group that did not receive ATIII.

Inclusion Criteria:

All sequential neonates (4-30 days of age) undergoing surgeries that require CPB at CHW are eligible to be included in the study.

Exclusion Criteria:

Patients with a prior operation utilizing CPB, weight less than 2 kilograms, prematurity less than 37 weeks estimated gestational age, previously diagnosed pro-thrombotic or hemorrhagic disorder, known intracranial hemorrhage, prior ATIII supplementation, and prior therapeutic anticoagulant use.

Protocol:

After informed consent, patients will be risk stratified into two groups based on whether the planned surgery will result in a cyanotic or acyanotic palliation. The patients in these two groups will then be randomized to either the ATIII group or the placebo group. A preoperative ATIII blood level will be obtained. This level will guide the dosing of ATIII or placebo, as neonatal congenital heart disease patients have variable baseline ATIII levels. The dose of ATIII or placebo will be determined by the following formula, in order to obtain ATIII blood levels similar to adults and older children (1.0 U/mL):

ATIII dose given to patient (U) = [(1.0 U/mL - patient's measured ATIII concentration in U/mL) X weight (kg) X 80 mL/kg]

This formula is derived by taking into account the volume of distribution of ATIII in the patient's blood volume. 80 mL/kg is an average blood volume for an infant. 1.0 U/ml is the normal level for older children and adults, and the target level we are trying to achieve. The patient's baseline level is subtracted from the target level to determine the relative ATIII deficiency in terms of U/mL. That amount is then multiplied by the estimated blood volume of 80 mL/kg and the patient's weight in kg to determine an ATIII dose in Units. The CHW pharmacy will use the above formula to obtain the appropriate dose of ATIII or placebo for each patient. ATIII or placebo will be administered after induction of general anesthesia and prior to administration of heparin and initiation of CPB. All treating physicians and study personal except for the preparing pharmacist will be blinded.

Heparin management during CPB will be accomplished according to the current standard practice at CHW. Anticoagulation during bypass will be monitored and titrated by use of the Medtronic Hepcon® HMS Plus Hemostasis Management System. A 3mL sample of the patient's blood is drawn pre-incision, after ATIII or placebo dosing, and is used by the HMS device to determine the in vitro individual response to heparin. A patient-specific heparin dose of between 300 and 800 units/kg will be administered before initiation of CPB, with the appropriate level of anticoagulation maintained at a minimum activated clotting time (ACT) of 480 seconds. The level of anticoagulation will be measured every half hour during CPB, with additional doses of heparin periodically administered as dictated by the HMS System measurements. At the completion of CPB, the heparin will be reversed with a patient-specific protamine dose, as calculated by the HMS System. Repeat measurements of ACT and heparin levels with the HMS device will be done after protamine administration to insure adequate reversal of the heparin effect.

ATIII levels will be measured within 5-10 minutes after administration (prior to start of CPB), within 30 minutes of start of CPB, just prior to discontinuation of CPB (prior to protamine dosing), and upon admission to the ICU. These levels will be kept blinded to all treating physicians and study personal.

An additional 2 mL of blood will be drawn at each time an ATIII level is obtained (total of 10 mL) to measure markers of activation of the coagulation and inflammatory systems, in order to better characterize the derangements in this patient population over time. We intend to use these results to develop future studies.

Intraoperative blood loss while on the CPB machine will be collected and placed back in the CPB circuit as per standard practice at CHW. Blood loss (mL/kg) will be determined intraoperatively from 10 minutes after protamine administration until admission to the intensive care unit (ICU). Chest tube output will then be recorded as a measure of blood loss for the first 24 hours after admission to the ICU.

After admission to the ICU, a transfusion protocol will then be used to ensure common indications for blood product replacement. Patients will be transfused with pRBC (10-15 mL/kg) if their hematocrit is less than 42% (higher target for evidence of inadequate oxygen delivery such as low SvO2, decreased cerebral NIRS, rising lactate, etc.). This protocol is consistent with our current standard practice at CHW.

If the bedside clinician decides a transfusion is/is not indicated outside of these guidelines, it will be recorded as a protocol variation and will be analyzed inclusively and separately. Volume of whole blood transfused will be multiplied by 0.5, as the concentration of red blood cells in whole blood is about 0.5 times the concentration present in packed red blood cells.

Additional serum blood samples will be drawn preoperatively and postoperatively (on the day the last invasive line is in place or 28 days postoperatively whichever is first) to determine antibody formation to recombinant antithrombin and goat milk proteins as a measure of safety of the specific ATIII product used.

Data Collection, Analysis, and Power Calculation:

Data will be recorded on a standardized data collection forms and stored in a RedCap data base which allows for menu driven options, inbuilt checks and generation of reports.

Safety (Aim 1): We hypothesize that measurements of safety in the experimental group will be the same or less than in the placebo controls We will record the mortality rate, incidence of extracorporeal membrane oxygenation (ECMO) support within 24 hours postoperatively, incidence of mediastinal exploration for bleeding and other indications within 24 hours postoperatively, incidence of thrombotic disease at discharge (ultrasound or other radiographic evidence if obtained for routine patient care), incidence of intracranial hemorrhage (ultrasound or computed tomography if obtained for routine patient care), days to delayed sternal closure, days to cessation of mechanical ventilation, and days to hospital discharge in the experimental and control groups. We will compare these data using a chi-square for categorical data, a t-test for continuous data, and Kaplan Meir curves with a Wilcoxon rank sum test for censored data. We will also compare serum samples at baseline and postoperatively for antibody formation to recombinant antithrombin or goat milk proteins. An internal data safety monitoring board (DSMB) will be in place to review the safety of the study after every patient for the first five, and then after every subsequent five patients. In addition, the DSMB will convene to review any serious adverse events potentially related to ATryn administration. A serious adverse event will be defined as death, intracranial hemorrhage, or >60 ml/kg/day in pRBC transfusion volume and/or 120 ml/kg/day of chest tube output (2 standard deviations above the mean in historical controls). At all points when the DSMB is planned to meet, the study will be placed on temporary hold, and no subsequent patients will be enrolled until after the DSMB convenes. If the DSMB concludes that ATryn administration contributed to a serious adverse event, or that the rates of safety measures described above are significantly worse in the ATryn-treated group at the time of a review, the study will be stopped.

Feasibility (Aim 1): We hypothesize that recruitment will be at a rate of 5 enrolled patients per month.

During the course of this project, the number of subjects approached for consent, the number consented, and difficulties in measurement (including unobtainable measures) will be summarized overall and by demographics. Associations will be investigated with scatter plots, Loess smooth curves, and Pearson correlation coefficients.

ATIII Pharmacokinetics (Aim 2): ATIII levels measured within 5-10 minutes after administration (prior to start of CPB), within 30 minutes of start of CPB, just prior to discontinuation of CPB (prior to protamine dosing), and upon admission to the ICU will be assessed to determine if the single dose of ATIII sustained normal ATIII levels in the experimental group throughout these time periods, and will be compared to placebo control patients. If any ATIII level is above 1.2 (20% higher than anticipated based on dose calculation) at the time of a review by the DSMB, the study will be placed on temporary hold in order to review the dose calculation protocol.

Postoperative Blood Loss and pRBC Transfusion Volume (Aim 3): Our primary efficacy hypothesis for this study is that blood loss and pRBC transfusion volumes will be less than placebo. Blood loss will be measured in terms of volumes (mL/kg) of blood loss and chest tube output from 10 minutes after protamine administration to 24 hours after ICU admission. If a patient requires re-exploration of the chest in the first 24 hours postoperatively, the volume of chest tube output for the duration of exploration will be recorded as a time-weighted average equal to the chest tube loss for the 2 hours prior to and 2 hours after the exploration. Volumes (mL/kg) of packed red blood cells and 0.5 X volume (mL/kg) of whole blood transfused from 10 minutes after protamine administration to 24 hours after ICU admission will be recorded. Patients who require ECMO within the first 24 hours postoperatively will be analyzed separately, as this is a known risk factor of increased bleeding and transfusion support. We will compare the blood loss and pRBC transfusion volumes in the two groups using a t-test or a Mann Whitney test. Further, we will allow for demographics such as sex and race, using a regression model with blood loss or pRBC volume as the outcome and group, and demographics as the independent variables.

Power analysis: Since there are two primary outcomes of blood loss volume and pRBC transfusion volume, we will use a Bonferroni adjustment and an alpha of 0.05/2= 0.025. With 30 patients in the experimental group and 30 controls, we will have at least 80% power to detect a difference of 0.81 standard deviations.

ELIGIBILITY:
Inclusion Criteria:

all sequential neonates (4 - 30 days of age) undergoing surgery requiring cardiopulmonary bypass are eligible to be included in the study.

Exclusion Criteria:

* prior operation utilizing cardiopulmonary bypass
* weight less than 2 kilograms
* prematurity less than 37 weeks estimated gestational age
* previously diagnosed pro-thrombotic or hemorrhagic disorder
* known intracranial hemorrhage
* prior ATIII supplementation
* prior therapeutic anticoagulant use
* known hypersensitivity to goat and goat milk proteins.

Ages: 4 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Measurements of safety will be same or less than placebo controls. | Hospital Discharge
  Mortality rate, incidence of ECMO support within 24 hours postoperatively, incidence of mediastinal exploration within 24 hours postoperatively, incidence of thrombotic disease at discharge (ultrasound or other radiographic evidence if obtained for routine patient care), incidence of intracranial hemorrhage (ultrasound or computed tomography if obtained for routine patient care), days to delayed sternal closure, days to cessation of mechanical ventilation, and days to hospital discharge in the experimental and control groups.

SECONDARY OUTCOMES:
Postoperative blood loss | 24 hours postoperatively
  Blood loss will be volumes (mL/kg) of blood loss and chest tube output from 10 minutes after protamine administration to 24 hours after ICU admission. We will compare this data to placebo controls.
Postoperative pRBC transfusion volume | 24 hours postoperatively
  Transfusion will be volumes (mL/kg) of pRBC transfuion and 0.5 times volumes (mL/kg) of whole blood transfusion from 10 minutes after protamine administration to 24 hours after ICU admission. We will compare this data to placebo controls.
ATIII pharmacokinetics | 24 hours postoperatively
  ATIII levels drawn preoperatively, within 30 minutes after administration (prior to start of CPB), within 30 minutes of start of CPB, just prior to discontinuation of CPB, and upon admission to the ICU will be assessed to determine if the single dose of ATIII sustained normal ATIII levels in the experimental group throughout these time periods.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Niebler, M.D., Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Murphy GJ, Reeves BC, Rogers CA, Rizvi SI, Culliford L, Angelini GD. Increased mortality, postoperative morbidity, and cost after red blood cell transfusion in patients having cardiac surgery. Circulation. 2007 Nov 27;116(22):2544-52. doi: 10.1161/CIRCULATIONAHA.107.698977. Epub 2007 Nov 12. PMID 17998460
- [Background] Engoren MC, Habib RH, Zacharias A, Schwann TA, Riordan CJ, Durham SJ. Effect of blood transfusion on long-term survival after cardiac operation. Ann Thorac Surg. 2002 Oct;74(4):1180-6. doi: 10.1016/s0003-4975(02)03766-9. PMID 12400765
- [Background] Spiess BD, Royston D, Levy JH, Fitch J, Dietrich W, Body S, Murkin J, Nadel A. Platelet transfusions during coronary artery bypass graft surgery are associated with serious adverse outcomes. Transfusion. 2004 Aug;44(8):1143-8. doi: 10.1111/j.1537-2995.2004.03322.x. PMID 15265117
- [Background] Chambers LA, Cohen DM, Davis JT. Transfusion patterns in pediatric open heart surgery. Transfusion. 1996 Feb;36(2):150-4. doi: 10.1046/j.1537-2995.1996.36296181928.x. PMID 8614966
- [Background] Petaja J, Lundstrom U, Leijala M, Peltola K, Siimes MA. Bleeding and use of blood products after heart operations in infants. J Thorac Cardiovasc Surg. 1995 Mar;109(3):524-9. doi: 10.1016/S0022-5223(95)70284-9. PMID 7877314
- [Background] Evans DA, Holder RL, Brawn WJ, Sethia B. Post-operative blood loss following cardio-pulmonary bypass in children. Eur J Cardiothorac Surg. 1994;8(1):25-9. doi: 10.1016/1010-7940(94)90128-7. PMID 8136165
- [Background] Bick RL. Alterations of hemostasis associated with cardiopulmonary bypass: pathophysiology, prevention, diagnosis, and management. Semin Thromb Hemost. 1976 Oct;3(2):59-82. doi: 10.1055/s-0028-1086129. PMID 798278
- [Background] Rosenberg RD. Biochemistry of heparin antithrombin interactions, and the physiologic role of this natural anticoagulant mechanism. Am J Med. 1989 Sep 11;87(3B):2S-9S. doi: 10.1016/0002-9343(89)80523-6. PMID 2679066
- [Background] Villaneuva GB, Danishefsky I. Evidence for a heparin-induced conformational change on antithrombin III. Biochem Biophys Res Commun. 1977 Jan 24;74(2):803-9. doi: 10.1016/0006-291x(77)90374-6. No abstract available. PMID 836327
- [Background] Despotis GJ, Levine V, Joist JH, Joiner-Maier D, Spitznagel E. Antithrombin III during cardiac surgery: effect on response of activated clotting time to heparin and relationship to markers of hemostatic activation. Anesth Analg. 1997 Sep;85(3):498-506. doi: 10.1097/00000539-199709000-00005. PMID 9296400
- [Background] Andrew M, Paes B, Milner R, Johnston M, Mitchell L, Tollefsen DM, Castle V, Powers P. Development of the human coagulation system in the healthy premature infant. Blood. 1988 Nov;72(5):1651-7. PMID 3179444
- [Background] Odegard KC, Zurakowski D, Hornykewycz S, DiNardo JA, Castro RA, Neufeld EJ, Laussen PC. Evaluation of the coagulation system in children with two-ventricle congenital heart disease. Ann Thorac Surg. 2007 May;83(5):1797-803. doi: 10.1016/j.athoracsur.2006.12.030. PMID 17462402
- [Background] Hakacova N, Laluhova-Striezencova Z, Zahorec M. Disturbances of coagulation in neonates with functionally univentricular physiology prior to the first stage of surgical reconstruction. Cardiol Young. 2008 Aug;18(4):397-401. doi: 10.1017/S1047951108002400. Epub 2008 Jun 18. PMID 18559135
- [Background] Odegard KC, Zurakowski D, DiNardo JA, Castro RA, McGowan FX Jr, Neufeld EJ, Laussen PC. Prospective longitudinal study of coagulation profiles in children with hypoplastic left heart syndrome from stage I through Fontan completion. J Thorac Cardiovasc Surg. 2009 Apr;137(4):934-41. doi: 10.1016/j.jtcvs.2008.09.031. Epub 2009 Feb 23. PMID 19327521
- [Background] Avidan MS, Levy JH, Scholz J, Delphin E, Rosseel PM, Howie MB, Gratz I, Bush CR, Skubas N, Aldea GS, Licina M, Bonfiglio LJ, Kajdasz DK, Ott E, Despotis GJ. A phase III, double-blind, placebo-controlled, multicenter study on the efficacy of recombinant human antithrombin in heparin-resistant patients scheduled to undergo cardiac surgery necessitating cardiopulmonary bypass. Anesthesiology. 2005 Feb;102(2):276-84. doi: 10.1097/00000542-200502000-00007. PMID 15681940
- [Background] Avidan MS, Levy JH, van Aken H, Feneck RO, Latimer RD, Ott E, Martin E, Birnbaum DE, Bonfiglio LJ, Kajdasz DK, Despotis GJ. Recombinant human antithrombin III restores heparin responsiveness and decreases activation of coagulation in heparin-resistant patients during cardiopulmonary bypass. J Thorac Cardiovasc Surg. 2005 Jul;130(1):107-13. doi: 10.1016/j.jtcvs.2004.10.045. PMID 15999048
- [Background] Koster A, Chew D, Kuebler W, Habazettl H, Hetzer R, Kuppe H. High antithrombin III levels attenuate hemostatic activation and leukocyte activation during cardiopulmonary bypass. J Thorac Cardiovasc Surg. 2003 Sep;126(3):906-7. doi: 10.1016/s0022-5223(03)00392-1. No abstract available. PMID 14502192
- [Background] Lemmer JH Jr, Despotis GJ. Antithrombin III concentrate to treat heparin resistance in patients undergoing cardiac surgery. J Thorac Cardiovasc Surg. 2002 Feb;123(2):213-7. doi: 10.1067/mtc.2002.119060. PMID 11828278
- [Background] Rinder CS, Rinder HM, Smith MJ, Fitch JC, Tracey JB, Chandler WL, Rollins SA, Smith BR. Antithrombin reduces monocyte and neutrophil CD11b up regulation in addition to blocking platelet activation during extracorporeal circulation. Transfusion. 2006 Jul;46(7):1130-7. doi: 10.1111/j.1537-2995.2006.00861.x. PMID 16836559
- [Background] Jaggers J, Lawson JH. Coagulopathy and inflammation in neonatal heart surgery: mechanisms and strategies. Ann Thorac Surg. 2006 Jun;81(6):S2360-6. doi: 10.1016/j.athoracsur.2006.02.072. No abstract available. PMID 16731104
- [Background] Agati S, Ciccarello G, Salvo D, Turla G, Undar A, Mignosa C. Use of a novel anticoagulation strategy during ECMO in a pediatric population: single-center experience. ASAIO J. 2006 Sep-Oct;52(5):513-6. doi: 10.1097/01.mat.0000242596.92625.a0. PMID 16966848